CLINICAL TRIAL: NCT00699335
Title: Efficacy of Matrifen® in Patients Older Than 18 Years With Severe, Chronic Pain Including Quality of Life Questionnaire
Brief Title: Matrifen® for Therapy of Severe Chronic Pain®
Acronym: Matrix LQ
Status: Completed | Type: Observational
Sponsor: Nycomed (Industry)
Responsible Party: Medical Responsible, Nycomed Deutschland GmbH
Other Study IDs: Matrix LQ, FT-1300-028
Record Dates: First submitted 2008-06-17; First posted 2008-06-18 (Estimated); Results first posted 2010-08-12 (Estimated); Last update posted 2012-05-08 (Estimated); Status verified 2012-05

CONDITIONS: Severe Chronic Pain
Keywords: pain; fentanyl; transdermal patch
MeSH Terms: conditions — Chronic Pain; Pain | interventions — Fentanyl

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Drug: Fentanyl — Fentanyl transdermal patch. This was an observational study - therefore, the physician decided about dosage according to individual needs

SUMMARY:
The aim of the study was to evaluate the efficacy and safety of Matrifen® in patients with severe and chronic pain who could only be sufficiently treated with opioid analgetics (WHO class 3).

ELIGIBILITY:
Main inclusion criteria:

* Outpatients with severe, chronic pain

Main exclusion criteria:

* Hypersensitivity to fentanyl
* Co-administration of monoamineoxidase-inhibitors
* Pregnancy
* Respiratory depression
* Chronic obstructive pulmonary disease (COPD)
* Drug abuse
* Impairment of CNS functions
* Other criteria as defined in the Summary of Product Characteristics (Chapter 4.3)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Outpatients
Sampling Method: Non-Probability Sample
Enrollment: 5308 (Actual)
Dates: Start 2008-06; Primary Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Thomas D. Bethke, MD, MBA, Study Director — Nycomed Deutschland GmbH, 78467 Konstanz, Germany
Locations (888):
- Germany (888):
  - Nycomed Deutschland GmbH, Aalen
  - Nycomed Deutschland GmbH, Abensberg
  - Nycomed Deutschland GmbH, Adelebsen
  - Nycomed Deutschland GmbH, Ahaus
  - Nycomed Deutschland GmbH, Ahlen
  - Nycomed Deutschland GmbH, Ahrensburg
  - Nycomed Deutschland GmbH, Albstadt
  - Nycomed Deutschland GmbH, Aldenhoven
  - Nycomed Deutschland GmbH, Alfeld
  - Nycomed Deutschland GmbH, Alfhausen
  - Nycomed Deutschland GmbH, Allersberg
  - Nycomed Deutschland GmbH, Alsfeld
  - Nycomed Deutschland GmbH, Altdorf
  - Nycomed Deutschland GmbH, Altenburg
  - Nycomed Deutschland GmbH, Altenstadt
  - Nycomed Deutschland GmbH, Althengstett
  - Nycomed Deutschland GmbH, Altlußheim
  - Nycomed Deutschland GmbH, Alzenau in Unterfranken
  - Nycomed Deutschland GmbH, Angermünde
  - Nycomed Deutschland GmbH, Annweiler am Trifels
  - Nycomed Deutschland GmbH, Ansbach
  - Nycomed Deutschland GmbH, Apolda
  - Nycomed Deutschland GmbH, Arnsberg
  - Nycomed Deutschland GmbH, Arnstadt
  - Nycomed Deutschland GmbH, Ascheberg
  - Nycomed Deutschland GmbH, Aschendorf
  - Nycomed Deutschland GmbH, Aschersleben
  - Nycomed Deutschland GmbH, Asslar-Werdorf
  - Nycomed Deutschland GmbH, Attendorn
  - Nycomed Deutschland GmbH, Attenkirchen
  - Nycomed Deutschland GmbH, Aue
  - Nycomed Deutschland GmbH, Auerbach
  - Nycomed Deutschland GmbH, Augsburg
  - Nycomed Deutschland GmbH, Augustdorf
  - Nycomed Deutschland GmbH, Aumühle
  - Nycomed Deutschland GmbH, Babenhausen
  - Nycomed Deutschland GmbH, Backnang
  - Nycomed Deutschland GmbH, Bad Arolsen
  - Nycomed Deutschland GmbH, Bad Bederkesa
  - Nycomed Deutschland GmbH, Bad Berka
  - Nycomed Deutschland GmbH, Bad Bevensen
  - Nycomed Deutschland GmbH, Bad Bramstedt
  - Nycomed Deutschland GmbH, Bad Düben
  - Nycomed Deutschland GmbH, Bad Dürkheim
  - Nycomed Deutschland GmbH, Bad Dürrenberg
  - Nycomed Deutschland GmbH, Bad Dürrheim
  - Nycomed Deutschland GmbH, Bad Eilsen
  - Nycomed Deutschland GmbH, Bad Essen
  - Nycomed Deutschland GmbH, Bad Frankenhausen
  - Nycomed Deutschland GmbH, Bad Homburg
  - Nycomed Deutschland GmbH, Bad Klosterlausnitz
  - Nycomed Deutschland GmbH, Bad Kreuznach
  - Nycomed Deutschland GmbH, Bad Krozingen
  - Nycomed Deutschland GmbH, Bad Langensalza
  - Nycomed Deutschland GmbH, Bad Lausick
  - Nycomed Deutschland GmbH, Bad Lauterberg im Harz
  - Nycomed Deutschland GmbH, Bad Liebenwerda
  - Nycomed Deutschland GmbH, Bad Nauheim
  - Nycomed Deutschland GmbH, Bad Neuenahr-Ahrweiler
  - Nycomed Deutschland GmbH, Bad Oeynhausen
  - Nycomed Deutschland GmbH, Bad Oldesloe
  - Nycomed Deutschland GmbH, Bad Salzuflen
  - Nycomed Deutschland GmbH, Bad Salzungen
  - Nycomed Deutschland GmbH, Bad Schandau
  - Nycomed Deutschland GmbH, Bad Schwalbach
  - Nycomed Deutschland GmbH, Bad Segeberg
  - Nycomed Deutschland GmbH, Bad Tennstedt
  - Nycomed Deutschland GmbH, Bad Tölz
  - Nycomed Deutschland GmbH, Bad Wilsnack
  - Nycomed Deutschland GmbH, Bad Windsheim
  - Nycomed Deutschland GmbH, Bad Wörishofen
  - Nycomed Deutschland GmbH, Badel
  - Nycomed Deutschland GmbH, Baden-Baden
  - Nycomed Deutschland GmbH, Badenhausen
  - Nycomed Deutschland GmbH, Badersleben
  - Nycomed Deutschland GmbH, Bahrdorf
  - Nycomed Deutschland GmbH, Bakum
  - Nycomed Deutschland GmbH, Balingen
  - Nycomed Deutschland GmbH, Ballrechten-Dottingen
  - Nycomed Deutschland GmbH, Bamberg
  - Nycomed Deutschland GmbH, Bautzen
  - Nycomed Deutschland GmbH, Bayreuth
  - Nycomed Deutschland GmbH, Beckum
  - Nycomed Deutschland GmbH, Berching
  - Nycomed Deutschland GmbH, Bergfelde
  - Nycomed Deutschland GmbH, Bergisch Gladbach
  - Nycomed Deutschland GmbH, Bergkamen
  - Nycomed Deutschland GmbH, Bergrheinfeld
  - Nycomed Deutschland GmbH, Berlin
  - Nycomed Deutschland GmbH, Bernau
  - Nycomed Deutschland GmbH, Bernburg
  - Nycomed Deutschland GmbH, Berne
  - Nycomed Deutschland GmbH, Bernsbach
  - Nycomed Deutschland GmbH, Beselich
  - Nycomed Deutschland GmbH, Beucha
  - Nycomed Deutschland GmbH, Beverungen
  - Nycomed Deutschland GmbH, Biberach
  - Nycomed Deutschland GmbH, Bielefeld
  - Nycomed Deutschland GmbH, Bietigheim-Bissingen
  - Nycomed Deutschland GmbH, Bilzingsleben
  - Nycomed Deutschland GmbH, Bingen
  - Nycomed Deutschland GmbH, Bisingen
  - Nycomed Deutschland GmbH, Bitterfeld-Wolfen
  - Nycomed Deutschland GmbH, Blankenfelde-Mahlow
  - Nycomed Deutschland GmbH, Blankenhain
  - Nycomed Deutschland GmbH, Blieskastel
  - Nycomed Deutschland GmbH, Bobritzsch
  - Nycomed Deutschland GmbH, Bocholt
  - Nycomed Deutschland GmbH, Bochum
  - Nycomed Deutschland GmbH, Bodenwerder
  - Nycomed Deutschland GmbH, Bonndorf
  - Nycomed Deutschland GmbH, Borna
  - Nycomed Deutschland GmbH, Bottrop
  - Nycomed Deutschland GmbH, Boxberg
  - Nycomed Deutschland GmbH, Böblingen
  - Nycomed Deutschland GmbH, Böhlen
  - Nycomed Deutschland GmbH, Brake
  - Nycomed Deutschland GmbH, Brakel
  - Nycomed Deutschland GmbH, Bramsche
  - Nycomed Deutschland GmbH, Brand-Erbisdorf
  - Nycomed Deutschland GmbH, Braunsbedra
  - Nycomed Deutschland GmbH, Braunschweig
  - Nycomed Deutschland GmbH, Bredstedt
  - Nycomed Deutschland GmbH, Breidenbach
  - Nycomed Deutschland GmbH, Breitenbrunn
  - Nycomed Deutschland GmbH, Bremen
  - Nycomed Deutschland GmbH, Bremerhaven
  - Nycomed Deutschland GmbH, Bremervörde
  - Nycomed Deutschland GmbH, Brilon
  - Nycomed Deutschland GmbH, Bruchsal
  - Nycomed Deutschland GmbH, Bruck
  - Nycomed Deutschland GmbH, Brüel
  - Nycomed Deutschland GmbH, Burg
  - Nycomed Deutschland GmbH, Burgbrohl
  - Nycomed Deutschland GmbH, Burgdorf, Hanover
  - Nycomed Deutschland GmbH, Burgstädt
  - Nycomed Deutschland GmbH, Burkardroth
  - Nycomed Deutschland GmbH, Burkhardtsdorf
  - Nycomed Deutschland GmbH, Burscheid
  - Nycomed Deutschland GmbH, Büchen
  - Nycomed Deutschland GmbH, Büchenbach
  - Nycomed Deutschland GmbH, Bückeburg
  - Nycomed Deutschland GmbH, Bühl-Altschweier
  - Nycomed Deutschland GmbH, Bühlertann
  - Nycomed Deutschland GmbH, Castrop-Rauxel
  - Nycomed Deutschland GmbH, Celle
  - Nycomed Deutschland GmbH, Chemnitz
  - Nycomed Deutschland GmbH, Clausthal-Zellerfeld
  - Nycomed Deutschland GmbH, Claußnitz
  - Nycomed Deutschland GmbH, Clenze
  - Nycomed Deutschland GmbH, Cloppenburg
  - Nycomed Deutschland GmbH, Coburg
  - Nycomed Deutschland GmbH, Cochem
  - Nycomed Deutschland GmbH, Coesfeld
  - Nycomed Deutschland GmbH, Cologne
  - Nycomed Deutschland GmbH, Coswig
  - Nycomed Deutschland GmbH, Cottbus
  - Nycomed Deutschland GmbH, Cölbe
  - Nycomed Deutschland GmbH, Crawinkel
  - Nycomed Deutschland GmbH, Crimmitschau
  - Nycomed Deutschland GmbH, Crivitz
  - Nycomed Deutschland GmbH, Crostwitz
  - Nycomed Deutschland GmbH, Cuxhaven
  - Nycomed Deutschland GmbH, Cuxhaven-Altenwalde
  - Nycomed Deutschland GmbH, Dachau
  - Nycomed Deutschland GmbH, Dahlwitz-Hoppegarten
  - Nycomed Deutschland GmbH, Darmstadt
  - Nycomed Deutschland GmbH, Dassel
  - Nycomed Deutschland GmbH, Dautphetal
  - Nycomed Deutschland GmbH, Deggendorf
  - Nycomed Deutschland GmbH, Deggingen
  - Nycomed Deutschland GmbH, Delitzsch
  - Nycomed Deutschland GmbH, Denzlingen
  - Nycomed Deutschland GmbH, Dessau
  - Nycomed Deutschland GmbH, Detmold
  - Nycomed Deutschland GmbH, Dettenheim
  - Nycomed Deutschland GmbH, Dettmannsdorf-Kölzow
  - Nycomed Deutschland GmbH, Diedorf
  - Nycomed Deutschland GmbH, Diepholz
  - Nycomed Deutschland GmbH, Dillingen
  - Nycomed Deutschland GmbH, Dillingen-Diefflen
  - Nycomed Deutschland GmbH, Dinkelsbühl
  - Nycomed Deutschland GmbH, Dogern
  - Nycomed Deutschland GmbH, Dorsten
  - Nycomed Deutschland GmbH, Dortmund
  - Nycomed Deutschland GmbH, Döbeln
  - Nycomed Deutschland GmbH, Dörentrup
  - Nycomed Deutschland GmbH, Dörpen
  - Nycomed Deutschland GmbH, Dörzbach
  - Nycomed Deutschland GmbH, Dreieich
  - Nycomed Deutschland GmbH, Dresden
  - Nycomed Deutschland GmbH, Driedorf
  - Nycomed Deutschland GmbH, Duisburg
  - Nycomed Deutschland GmbH, Durach
  - Nycomed Deutschland GmbH, Durmersheim
  - Nycomed Deutschland GmbH, Düsseldorf
  - Nycomed Deutschland GmbH, Ebeleben
  - Nycomed Deutschland GmbH, Eberbach
  - Nycomed Deutschland GmbH, Ebersbach
  - Nycomed Deutschland GmbH, Eberswalde
  - Nycomed Deutschland GmbH, Eckernförde
  - Nycomed Deutschland GmbH, Eggenstein-Leopoldshafen
  - Nycomed Deutschland GmbH, Eggesin
  - Nycomed Deutschland GmbH, Ehingen
  - Nycomed Deutschland GmbH, Ehra-Lessien
  - Nycomed Deutschland GmbH, Ehrenkirchen-Kirchhofen
  - Nycomed Deutschland GmbH, Eibau
  - Nycomed Deutschland GmbH, Eimsheim
  - Nycomed Deutschland GmbH, Eisenach
  - Nycomed Deutschland GmbH, Eisenberg
  - Nycomed Deutschland GmbH, Eisenhüttenstadt
  - Nycomed Deutschland GmbH, Eisleben Lutherstadt
  - Nycomed Deutschland GmbH, Eiterfeld
  - Nycomed Deutschland GmbH, Ellhofen
  - Nycomed Deutschland GmbH, Ellwangen
  - Nycomed Deutschland GmbH, Elmshorn
  - Nycomed Deutschland GmbH, Elterlein
  - Nycomed Deutschland GmbH, Emleben
  - Nycomed Deutschland GmbH, Emsdetten
  - Nycomed Deutschland GmbH, Engelskirchen-Ründeroth
  - Nycomed Deutschland GmbH, Enkirch
  - Nycomed Deutschland GmbH, Eppingen
  - Nycomed Deutschland GmbH, Eppstein
  - Nycomed Deutschland GmbH, Eppstein/Ts.
  - Nycomed Deutschland GmbH, Erfurt
  - Nycomed Deutschland GmbH, Erkelenz
  - Nycomed Deutschland GmbH, Erlangen
  - Nycomed Deutschland GmbH, Eschelbronn
  - Nycomed Deutschland GmbH, Eschlkam
  - Nycomed Deutschland GmbH, Essen
  - Nycomed Deutschland GmbH, Faulbach
  - Nycomed Deutschland GmbH, Feldafing
  - Nycomed Deutschland GmbH, Felsberg
  - Nycomed Deutschland GmbH, Finsterwalde
  - Nycomed Deutschland GmbH, Flensburg
  - Nycomed Deutschland GmbH, Floh
  - Nycomed Deutschland GmbH, Flonheim
  - Nycomed Deutschland GmbH, Flörsheim-Dalsheim
  - Nycomed Deutschland GmbH, Forchheim
  - Nycomed Deutschland GmbH, Föhren
  - Nycomed Deutschland GmbH, Framersheim
  - Nycomed Deutschland GmbH, Frankenberg
  - Nycomed Deutschland GmbH, Frankenthal
  - Nycomed Deutschland GmbH, Frankfurt
  - Nycomed Deutschland GmbH, Freiberg
  - Nycomed Deutschland GmbH, Freiburg im Breisgau
  - Nycomed Deutschland GmbH, Freising
  - Nycomed Deutschland GmbH, Freyburg
  - Nycomed Deutschland GmbH, Friedeburg
  - Nycomed Deutschland GmbH, Friedrichsdorf
  - Nycomed Deutschland GmbH, Friedrichsthal
  - Nycomed Deutschland GmbH, Frohburg
  - Nycomed Deutschland GmbH, Furth im Wald
  - Nycomed Deutschland GmbH, Fürstenberg
  - Nycomed Deutschland GmbH, Fürstenstein
  - Nycomed Deutschland GmbH, Fürstenwalde
  - Nycomed Deutschland GmbH, Fürstenzell
  - Nycomed Deutschland GmbH, Fürth
  - Nycomed Deutschland GmbH, Gaggenau
  - Nycomed Deutschland GmbH, Gardelegen
  - Nycomed Deutschland GmbH, Garmisch-Partenkirchen
  - Nycomed Deutschland GmbH, Gebesee
  - Nycomed Deutschland GmbH, Geesthacht
  - Nycomed Deutschland GmbH, Geilenkirchen
  - Nycomed Deutschland GmbH, Geislingen
  - Nycomed Deutschland GmbH, Gelsenkirchen
  - Nycomed Deutschland GmbH, Gemünden
  - Nycomed Deutschland GmbH, Georgensgmünd
  - Nycomed Deutschland GmbH, Georgsmarienhütte
  - Nycomed Deutschland GmbH, Gera
  - Nycomed Deutschland GmbH, Gera-Lusan
  - Nycomed Deutschland GmbH, Gerbstedt
  - Nycomed Deutschland GmbH, Geretsried
  - Nycomed Deutschland GmbH, Germering
  - Nycomed Deutschland GmbH, Gernrode
  - Nycomed Deutschland GmbH, Gernsbach
  - Nycomed Deutschland GmbH, Gerzen
  - Nycomed Deutschland GmbH, Geyer
  - Nycomed Deutschland GmbH, Gladbeck
  - Nycomed Deutschland GmbH, Glaubitz
  - Nycomed Deutschland GmbH, Gleichen
  - Nycomed Deutschland GmbH, Goch
  - Nycomed Deutschland GmbH, Golzow
  - Nycomed Deutschland GmbH, Gomaringen
  - Nycomed Deutschland GmbH, Gommern
  - Nycomed Deutschland GmbH, Goslar
  - Nycomed Deutschland GmbH, Göllingen
  - Nycomed Deutschland GmbH, Göppingen
  - Nycomed Deutschland GmbH, Görlitz
  - Nycomed Deutschland GmbH, Göttingen
  - Nycomed Deutschland GmbH, Graben-Neudorf
  - Nycomed Deutschland GmbH, Gräfinau-Angstedt
  - Nycomed Deutschland GmbH, Grefrath
  - Nycomed Deutschland GmbH, Greiz
  - Nycomed Deutschland GmbH, Grimma
  - Nycomed Deutschland GmbH, Gronau
  - Nycomed Deutschland GmbH, Groß Ammensleben
  - Nycomed Deutschland GmbH, Groß Grönau
  - Nycomed Deutschland GmbH, Groß Wokern
  - Nycomed Deutschland GmbH, Großaitingen
  - Nycomed Deutschland GmbH, Großburschla
  - Nycomed Deutschland GmbH, Großefehn
  - Nycomed Deutschland GmbH, Großengottern
  - Nycomed Deutschland GmbH, Großerkmannsdorf
  - Nycomed Deutschland GmbH, Großharthau
  - Nycomed Deutschland GmbH, Großheirath-Rossach
  - Nycomed Deutschland GmbH, Großkorbetha
  - Nycomed Deutschland GmbH, Großlehna
  - Nycomed Deutschland GmbH, Gröden
  - Nycomed Deutschland GmbH, Grömitz
  - Nycomed Deutschland GmbH, Grundau
  - Nycomed Deutschland GmbH, Gundelsheim
  - Nycomed Deutschland GmbH, Gunzenhausen
  - Nycomed Deutschland GmbH, Güglingen
  - Nycomed Deutschland GmbH, Güsten
  - Nycomed Deutschland GmbH, Güster
  - Nycomed Deutschland GmbH, Hachenburg
  - Nycomed Deutschland GmbH, Hadamar
  - Nycomed Deutschland GmbH, Hagenow
  - Nycomed Deutschland GmbH, Haigerloch
  - Nycomed Deutschland GmbH, Halbe
  - Nycomed Deutschland GmbH, Halbendorf
  - Nycomed Deutschland GmbH, Halberstadt
  - Nycomed Deutschland GmbH, Haldensleben I
  - Nycomed Deutschland GmbH, Halle
  - Nycomed Deutschland GmbH, Hamburg
  - Nycomed Deutschland GmbH, Hamelin
  - Nycomed Deutschland GmbH, Hamm
  - Nycomed Deutschland GmbH, Hammelburg
  - Nycomed Deutschland GmbH, Hanau
  - Nycomed Deutschland GmbH, Hannoversch Münden
  - Nycomed Deutschland GmbH, Hanover
  - Nycomed Deutschland GmbH, Haren
  - Nycomed Deutschland GmbH, Harsewinkel
  - Nycomed Deutschland GmbH, Hartenstein
  - Nycomed Deutschland GmbH, Hartha
  - Nycomed Deutschland GmbH, Hattorf
  - Nycomed Deutschland GmbH, Haunsheim
  - Nycomed Deutschland GmbH, Hebertshausen
  - Nycomed Deutschland GmbH, Heckelberg-Brunow
  - Nycomed Deutschland GmbH, Heek
  - Nycomed Deutschland GmbH, Heidelberg
  - Nycomed Deutschland GmbH, Heilbad Heiligenstadt
  - Nycomed Deutschland GmbH, Heilbronn
  - Nycomed Deutschland GmbH, Heilsbronn
  - Nycomed Deutschland GmbH, Heinsdorfergrund
  - Nycomed Deutschland GmbH, Helmstedt
  - Nycomed Deutschland GmbH, Hemau
  - Nycomed Deutschland GmbH, Hemmoor
  - Nycomed Deutschland GmbH, Hennigsdorf
  - Nycomed Deutschland GmbH, Herborn
  - Nycomed Deutschland GmbH, Herbrechtingen
  - Nycomed Deutschland GmbH, Herbsleben
  - Nycomed Deutschland GmbH, Herne
  - Nycomed Deutschland GmbH, Heroldsberg
  - Nycomed Deutschland GmbH, Herrenberg
  - Nycomed Deutschland GmbH, Herrnhut
  - Nycomed Deutschland GmbH, Herxheim
  - Nycomed Deutschland GmbH, Hesel
  - Nycomed Deutschland GmbH, Hessen
  - Nycomed Deutschland GmbH, Hessisch Lichtenau
  - Nycomed Deutschland GmbH, Hettstedt
  - Nycomed Deutschland GmbH, Hildburghausen
  - Nycomed Deutschland GmbH, Hilden
  - Nycomed Deutschland GmbH, Hildesheim
  - Nycomed Deutschland GmbH, Hilzingen
  - Nycomed Deutschland GmbH, Hirschaid
  - Nycomed Deutschland GmbH, Hirschfelde
  - Nycomed Deutschland GmbH, Hockenheim
  - Nycomed Deutschland GmbH, Hofheim
  - Nycomed Deutschland GmbH, Hohenprießnitz
  - Nycomed Deutschland GmbH, Hollenstedt
  - Nycomed Deutschland GmbH, Hoyerswerda
  - Nycomed Deutschland GmbH, Höchheim
  - Nycomed Deutschland GmbH, Hörstel
  - Nycomed Deutschland GmbH, Höxter
  - Nycomed Deutschland GmbH, Husum
  - Nycomed Deutschland GmbH, Hückelhoven
  - Nycomed Deutschland GmbH, Hüllhorst
  - Nycomed Deutschland GmbH, Hüpstedt
  - Nycomed Deutschland GmbH, Hürth
  - Nycomed Deutschland GmbH, Ibbenbueren
  - Nycomed Deutschland GmbH, Ibbenbüren-Dickenberg
  - Nycomed Deutschland GmbH, Ilmenau
  - Nycomed Deutschland GmbH, Ilsenburg
  - Nycomed Deutschland GmbH, Ingelheim
  - Nycomed Deutschland GmbH, Ingolstadt
  - Nycomed Deutschland GmbH, Itzehoe
  - Nycomed Deutschland GmbH, Jarmen
  - Nycomed Deutschland GmbH, Jerichow
  - Nycomed Deutschland GmbH, Jessen
  - Nycomed Deutschland GmbH, Jettingen-Unterjettingen
  - Nycomed Deutschland GmbH, Joachimsthal
  - Nycomed Deutschland GmbH, Jockgrim
  - Nycomed Deutschland GmbH, Johanngeorgenstadt
  - Nycomed Deutschland GmbH, Jördenstorf
  - Nycomed Deutschland GmbH, Jübek
  - Nycomed Deutschland GmbH, Jüchen
  - Nycomed Deutschland GmbH, Jüterbog
  - Nycomed Deutschland GmbH, Kaisersesch
  - Nycomed Deutschland GmbH, Kaiserslautern
  - Nycomed Deutschland GmbH, Kalkar
  - Nycomed Deutschland GmbH, Kaltensundheim
  - Nycomed Deutschland GmbH, Kamen
  - Nycomed Deutschland GmbH, Kamenz
  - Nycomed Deutschland GmbH, Kandern
  - Nycomed Deutschland GmbH, Kappeln
  - Nycomed Deutschland GmbH, Karlsbad
  - Nycomed Deutschland GmbH, Karlsdorf-Neuthard
  - Nycomed Deutschland GmbH, Karlsruhe
  - Nycomed Deutschland GmbH, Karstädt
  - Nycomed Deutschland GmbH, Kassel
  - Nycomed Deutschland GmbH, Katzhütte
  - Nycomed Deutschland GmbH, Kaufbeuren
  - Nycomed Deutschland GmbH, Käbschütztal
  - Nycomed Deutschland GmbH, Kelkheim
  - Nycomed Deutschland GmbH, Keltern
  - Nycomed Deutschland GmbH, Kemnitz
  - Nycomed Deutschland GmbH, Kempen
  - Nycomed Deutschland GmbH, Kempenich
  - Nycomed Deutschland GmbH, Kempten
  - Nycomed Deutschland GmbH, Ketsch
  - Nycomed Deutschland GmbH, Kiel
  - Nycomed Deutschland GmbH, Kipfenberg
  - Nycomed Deutschland GmbH, Kirchberg
  - Nycomed Deutschland GmbH, Kirchehrenbach
  - Nycomed Deutschland GmbH, Kirchenlamitz
  - Nycomed Deutschland GmbH, Kirchheimbolanden
  - Nycomed Deutschland GmbH, Kirchzarten
  - Nycomed Deutschland GmbH, Kleve
  - Nycomed Deutschland GmbH, Klingenthal
  - Nycomed Deutschland GmbH, Kloster Lehnin
  - Nycomed Deutschland GmbH, Koblenz
  - Nycomed Deutschland GmbH, Kolbermoor
  - Nycomed Deutschland GmbH, Kornwestheim
  - Nycomed Deutschland GmbH, Koßdorf
  - Nycomed Deutschland GmbH, Köhra
  - Nycomed Deutschland GmbH, Köln-Höhenberg
  - Nycomed Deutschland GmbH, Königs Wusterhausen
  - Nycomed Deutschland GmbH, Königswartha
  - Nycomed Deutschland GmbH, Kösching
  - Nycomed Deutschland GmbH, Köthen
  - Nycomed Deutschland GmbH, Krauschwitz
  - Nycomed Deutschland GmbH, Krefeld
  - Nycomed Deutschland GmbH, Kreuztal
  - Nycomed Deutschland GmbH, Krippen
  - Nycomed Deutschland GmbH, Kronach
  - Nycomed Deutschland GmbH, Kronau
  - Nycomed Deutschland GmbH, Krumpa
  - Nycomed Deutschland GmbH, Kurort Seiffen
  - Nycomed Deutschland GmbH, Kühbach
  - Nycomed Deutschland GmbH, Küllstedt
  - Nycomed Deutschland GmbH, Laatzen
  - Nycomed Deutschland GmbH, Lahnau
  - Nycomed Deutschland GmbH, Lampertheim
  - Nycomed Deutschland GmbH, Lamstedt
  - Nycomed Deutschland GmbH, Landau
  - Nycomed Deutschland GmbH, Langelsheim
  - Nycomed Deutschland GmbH, Langenbrettach
  - Nycomed Deutschland GmbH, Langenfeld
  - Nycomed Deutschland GmbH, Langenhagen
  - Nycomed Deutschland GmbH, Lauf
  - Nycomed Deutschland GmbH, Laufenburg
  - Nycomed Deutschland GmbH, Lauingen
  - Nycomed Deutschland GmbH, Lebach
  - Nycomed Deutschland GmbH, Leer
  - Nycomed Deutschland GmbH, Leiblfing
  - Nycomed Deutschland GmbH, Leimen
  - Nycomed Deutschland GmbH, Leinefelde-Worbis
  - Nycomed Deutschland GmbH, Leinefelde
  - Nycomed Deutschland GmbH, Leipheim
  - Nycomed Deutschland GmbH, Leipzig
  - Nycomed Deutschland GmbH, Lemförde
  - Nycomed Deutschland GmbH, Lengefeld
  - Nycomed Deutschland GmbH, Lengerich
  - Nycomed Deutschland GmbH, Lensahn
  - Nycomed Deutschland GmbH, Leubnitz
  - Nycomed Deutschland GmbH, Leutkirch
  - Nycomed Deutschland GmbH, Leverkusen
  - Nycomed Deutschland GmbH, Leverkusen-Hitdorf
  - Nycomed Deutschland GmbH, Lichtenfels
  - Nycomed Deutschland GmbH, Lichtenstein
  - Nycomed Deutschland GmbH, Lilienthal
  - Nycomed Deutschland GmbH, Limburgerhof
  - Nycomed Deutschland GmbH, Lohfelden
  - Nycomed Deutschland GmbH, Lohsa
  - Nycomed Deutschland GmbH, Lommatzsch
  - Nycomed Deutschland GmbH, Lorch
  - Nycomed Deutschland GmbH, Löbau
  - Nycomed Deutschland GmbH, Löbejün
  - Nycomed Deutschland GmbH, Löhne
  - Nycomed Deutschland GmbH, Lubnjow
  - Nycomed Deutschland GmbH, Ludwigsburg
  - Nycomed Deutschland GmbH, Ludwigshafen
  - Nycomed Deutschland GmbH, Ludwigsstadt
  - Nycomed Deutschland GmbH, Lübeck
  - Nycomed Deutschland GmbH, Lüneburg
  - Nycomed Deutschland GmbH, Lünen
  - Nycomed Deutschland GmbH, Magdeburg
  - Nycomed Deutschland GmbH, Mainaschaff
  - Nycomed Deutschland GmbH, Mainz
  - Nycomed Deutschland GmbH, Malchin
  - Nycomed Deutschland GmbH, Malchow
  - Nycomed Deutschland GmbH, Mannheim
  - Nycomed Deutschland GmbH, Marburg
  - Nycomed Deutschland GmbH, Marienberg
  - Nycomed Deutschland GmbH, Marienheide
  - Nycomed Deutschland GmbH, Markkleeberg
  - Nycomed Deutschland GmbH, Meckenheim
  - Nycomed Deutschland GmbH, Meinhard
  - Nycomed Deutschland GmbH, Meißen
  - Nycomed Deutschland GmbH, Mellrichstadt
  - Nycomed Deutschland GmbH, Memmingen
  - Nycomed Deutschland GmbH, Menden
  - Nycomed Deutschland GmbH, Mendig
  - Nycomed Deutschland GmbH, Mengen
  - Nycomed Deutschland GmbH, Menteroda
  - Nycomed Deutschland GmbH, Merkendorf
  - Nycomed Deutschland GmbH, Merseburg
  - Nycomed Deutschland GmbH, Merzig
  - Nycomed Deutschland GmbH, Mettlach
  - Nycomed Deutschland GmbH, Metzingen
  - Nycomed Deutschland GmbH, Meuselwitz
  - Nycomed Deutschland GmbH, Mildstedt
  - Nycomed Deutschland GmbH, Mindelstetten
  - Nycomed Deutschland GmbH, Minden
  - Nycomed Deutschland GmbH, Mittelherwigsdorf
  - Nycomed Deutschland GmbH, Moers
  - Nycomed Deutschland GmbH, Monheim
  - Nycomed Deutschland GmbH, Monschau
  - Nycomed Deutschland GmbH, Montabaur
  - Nycomed Deutschland GmbH, Mosbach
  - Nycomed Deutschland GmbH, Mosbach-Lohrbach
  - Nycomed Deutschland GmbH, Möckern
  - Nycomed Deutschland GmbH, Möhlau
  - Nycomed Deutschland GmbH, Mölln
  - Nycomed Deutschland GmbH, Mönchengladbach
  - Nycomed Deutschland GmbH, Mühlberg
  - Nycomed Deutschland GmbH, Mühlenbeck
  - Nycomed Deutschland GmbH, Mühlhausen
  - Nycomed Deutschland GmbH, Mülheim
  - Nycomed Deutschland GmbH, Mülsen
  - Nycomed Deutschland GmbH, München
  - Nycomed Deutschland GmbH, Münster
  - Nycomed Deutschland GmbH, Münzenberg-Gambach
  - Nycomed Deutschland GmbH, Nassau
  - Nycomed Deutschland GmbH, Nastätten
  - Nycomed Deutschland GmbH, Nattheim
  - Nycomed Deutschland GmbH, Nauen
  - Nycomed Deutschland GmbH, Naumburg
  - Nycomed Deutschland GmbH, Neckarbischofsheim
  - Nycomed Deutschland GmbH, Neckargemünd
  - Nycomed Deutschland GmbH, Neckarsulm
  - Nycomed Deutschland GmbH, Nettersheim
  - Nycomed Deutschland GmbH, Netzschkau
  - Nycomed Deutschland GmbH, Neu Wulmstorf
  - Nycomed Deutschland GmbH, Neu-Anspach
  - Nycomed Deutschland GmbH, Neu-Isenburg
  - Nycomed Deutschland GmbH, Neubrandenburg
  - Nycomed Deutschland GmbH, Neudietendorf
  - Nycomed Deutschland GmbH, Neuenhagen
  - Nycomed Deutschland GmbH, Neuenkirchen-Vörden
  - Nycomed Deutschland GmbH, Neufahrn
  - Nycomed Deutschland GmbH, Neuhof
  - Nycomed Deutschland GmbH, Neukieritzsch
  - Nycomed Deutschland GmbH, Neukirch
  - Nycomed Deutschland GmbH, Neukirchen
  - Nycomed Deutschland GmbH, Neukirchen-Vluyn
  - Nycomed Deutschland GmbH, Neumünster
  - Nycomed Deutschland GmbH, Neunkirchen
  - Nycomed Deutschland GmbH, Neuruppin
  - Nycomed Deutschland GmbH, Neuseußlitz
  - Nycomed Deutschland GmbH, Neuss
  - Nycomed Deutschland GmbH, Neustadt
  - Nycomed Deutschland GmbH, Neustadt in Sachsen
  - Nycomed Deutschland GmbH, Nieder-Olm
  - Nycomed Deutschland GmbH, Niederlehme
  - Nycomed Deutschland GmbH, Niendorf
  - Nycomed Deutschland GmbH, Norderstedt
  - Nycomed Deutschland GmbH, Nordhausen
  - Nycomed Deutschland GmbH, Nordhorn
  - Nycomed Deutschland GmbH, Nordstemmen
  - Nycomed Deutschland GmbH, Nossen
  - Nycomed Deutschland GmbH, Nördlingen
  - Nycomed Deutschland GmbH, Nuremberg
  - Nycomed Deutschland GmbH, Obercunnersdorf
  - Nycomed Deutschland GmbH, Oberdorla
  - Nycomed Deutschland GmbH, Oberhausen
  - Nycomed Deutschland GmbH, Obertshausen
  - Nycomed Deutschland GmbH, Oberursel
  - Nycomed Deutschland GmbH, Oberursel/Ts. Oberstedten
  - Nycomed Deutschland GmbH, Ochtendung
  - Nycomed Deutschland GmbH, Oderwitz
  - Nycomed Deutschland GmbH, Oelsnitz
  - Nycomed Deutschland GmbH, Oer-Erkenschwick
  - Nycomed Deutschland GmbH, Oerel
  - Nycomed Deutschland GmbH, Offenburg
  - Nycomed Deutschland GmbH, Oftersheim
  - Nycomed Deutschland GmbH, Olbersdorf
  - Nycomed Deutschland GmbH, Oldenburg
  - Nycomed Deutschland GmbH, Oldendorf
  - Nycomed Deutschland GmbH, Olpe
  - Nycomed Deutschland GmbH, Oranienburg
  - Nycomed Deutschland GmbH, Oschatz
  - Nycomed Deutschland GmbH, Osloß
  - Nycomed Deutschland GmbH, Osnabrück
  - Nycomed Deutschland GmbH, Ostbevern
  - Nycomed Deutschland GmbH, Osterburg
  - Nycomed Deutschland GmbH, Osterode
  - Nycomed Deutschland GmbH, Ostrhauderfehn
  - Nycomed Deutschland GmbH, Ostseebad Kühlungsborn
  - Nycomed Deutschland GmbH, Ottendorf-Okrilla
  - Nycomed Deutschland GmbH, Otterndorf
  - Nycomed Deutschland GmbH, Ottersberg
  - Nycomed Deutschland GmbH, Overath
  - Nycomed Deutschland GmbH, Östringen
  - Nycomed Deutschland GmbH, Paderborn
  - Nycomed Deutschland GmbH, Panitzsch
  - Nycomed Deutschland GmbH, Panketal
  - Nycomed Deutschland GmbH, Panschwitz-Kuckau
  - Nycomed Deutschland GmbH, Papenburg
  - Nycomed Deutschland GmbH, Parchim
  - Nycomed Deutschland GmbH, Passau
  - Nycomed Deutschland GmbH, Passau/Hacklberg
  - Nycomed Deutschland GmbH, Peckelsheim
  - Nycomed Deutschland GmbH, Peine
  - Nycomed Deutschland GmbH, Penig
  - Nycomed Deutschland GmbH, Perleberg
  - Nycomed Deutschland GmbH, Petershagen
  - Nycomed Deutschland GmbH, Pfaffenhofen
  - Nycomed Deutschland GmbH, Pforzheim
  - Nycomed Deutschland GmbH, Pfullingen
  - Nycomed Deutschland GmbH, Pfungstadt
  - Nycomed Deutschland GmbH, Pilsting
  - Nycomed Deutschland GmbH, Pirmasens
  - Nycomed Deutschland GmbH, Plauen
  - Nycomed Deutschland GmbH, Plessa
  - Nycomed Deutschland GmbH, Plön
  - Nycomed Deutschland GmbH, Pohlheim
  - Nycomed Deutschland GmbH, Polch
  - Nycomed Deutschland GmbH, Porta Westfalica
  - Nycomed Deutschland GmbH, Potsdam
  - Nycomed Deutschland GmbH, Pößneck
  - Nycomed Deutschland GmbH, Prausitz
  - Nycomed Deutschland GmbH, Prösen
  - Nycomed Deutschland GmbH, Pulheim
  - Nycomed Deutschland GmbH, Pullach
  - Nycomed Deutschland GmbH, Pulsnitz
  - Nycomed Deutschland GmbH, Puschwitz
  - Nycomed Deutschland GmbH, Quedlinburg
  - Nycomed Deutschland GmbH, Rabenau
  - Nycomed Deutschland GmbH, Radebeul
  - Nycomed Deutschland GmbH, Radevormwald
  - Nycomed Deutschland GmbH, Rastede
  - Nycomed Deutschland GmbH, Regensburg
  - Nycomed Deutschland GmbH, Reichenbach
  - Nycomed Deutschland GmbH, Reinfeld
  - Nycomed Deutschland GmbH, Remagen
  - Nycomed Deutschland GmbH, Remchingen-Singen
  - Nycomed Deutschland GmbH, Remscheid
  - Nycomed Deutschland GmbH, Rendsburg
  - Nycomed Deutschland GmbH, Reutlingen
  - Nycomed Deutschland GmbH, Ribnitz-Damgarten
  - Nycomed Deutschland GmbH, Riedlingen
  - Nycomed Deutschland GmbH, Rippien
  - Nycomed Deutschland GmbH, Rodenbach
  - Nycomed Deutschland GmbH, Rodewisch
  - Nycomed Deutschland GmbH, Rohrbach
  - Nycomed Deutschland GmbH, Rosenfeld
  - Nycomed Deutschland GmbH, Rosengarten
  - Nycomed Deutschland GmbH, Rostock
  - Nycomed Deutschland GmbH, Rotenburg (Wümme)
  - Nycomed Deutschland GmbH, Rothenburg
  - Nycomed Deutschland GmbH, Rottenburg
  - Nycomed Deutschland GmbH, Rottleberode
  - Nycomed Deutschland GmbH, Roßtal
  - Nycomed Deutschland GmbH, Rödermark
  - Nycomed Deutschland GmbH, Röhrmoos
  - Nycomed Deutschland GmbH, Rösrath
  - Nycomed Deutschland GmbH, Rudolstadt
  - Nycomed Deutschland GmbH, Rülzheim
  - Nycomed Deutschland GmbH, Rüsselsheim am Main
  - Nycomed Deutschland GmbH, Saalburg-Ebersdorf
  - Nycomed Deutschland GmbH, Saalfeld
  - Nycomed Deutschland GmbH, Saarbrücken
  - Nycomed Deutschland GmbH, Saint Ingbert
  - Nycomed Deutschland GmbH, Salzgitter
  - Nycomed Deutschland GmbH, Salzkotten
  - Nycomed Deutschland GmbH, Salzmünde
  - Nycomed Deutschland GmbH, Sand
  - Nycomed Deutschland GmbH, Sandesneben
  - Nycomed Deutschland GmbH, Sangerhausen
  - Nycomed Deutschland GmbH, Sankt Leon-Rot
  - Nycomed Deutschland GmbH, Sarstedt
  - Nycomed Deutschland GmbH, Sayda
  - Nycomed Deutschland GmbH, Schellerten
  - Nycomed Deutschland GmbH, Scheßlitz
  - Nycomed Deutschland GmbH, Schladen
  - Nycomed Deutschland GmbH, Schleswig
  - Nycomed Deutschland GmbH, Schliersee-Neuhaus
  - Nycomed Deutschland GmbH, Schmalkalden
  - Nycomed Deutschland GmbH, Schneeberg
  - Nycomed Deutschland GmbH, Schonungen
  - Nycomed Deutschland GmbH, Schortens
  - Nycomed Deutschland GmbH, Schömberg
  - Nycomed Deutschland GmbH, Schönberg
  - Nycomed Deutschland GmbH, Schöneck
  - Nycomed Deutschland GmbH, Schönwalde
  - Nycomed Deutschland GmbH, Schriesheim
  - Nycomed Deutschland GmbH, Schwaan
  - Nycomed Deutschland GmbH, Schwabach
  - Nycomed Deutschland GmbH, Schwaig
  - Nycomed Deutschland GmbH, Schwalmstadt
  - Nycomed Deutschland GmbH, Schwandorf in Bayern
  - Nycomed Deutschland GmbH, Schwanewede
  - Nycomed Deutschland GmbH, Schwanstetten
  - Nycomed Deutschland GmbH, Schwarmstedt
  - Nycomed Deutschland GmbH, Schwarzenbruck
  - Nycomed Deutschland GmbH, Schwäbisch Gmünd
  - Nycomed Deutschland GmbH, Schwedt
  - Nycomed Deutschland GmbH, Schweinitz
  - Nycomed Deutschland GmbH, Schwerin
  - Nycomed Deutschland GmbH, Schwetzingen
  - Nycomed Deutschland GmbH, Seeheilbad Graal-Müritz
  - Nycomed Deutschland GmbH, Seeheim-Jugenheim
  - Nycomed Deutschland GmbH, Sickte
  - Nycomed Deutschland GmbH, Siegen
  - Nycomed Deutschland GmbH, Silberhausen
  - Nycomed Deutschland GmbH, Simmertal
  - Nycomed Deutschland GmbH, Sindelfingen
  - Nycomed Deutschland GmbH, Singen
  - Nycomed Deutschland GmbH, Solingen
  - Nycomed Deutschland GmbH, Sonneberg
  - Nycomed Deutschland GmbH, Sonsbeck
  - Nycomed Deutschland GmbH, Sömmerda
  - Nycomed Deutschland GmbH, Spalt
  - Nycomed Deutschland GmbH, Speichersdorf
  - Nycomed Deutschland GmbH, Speyer
  - Nycomed Deutschland GmbH, Spremberg
  - Nycomed Deutschland GmbH, Springe
  - Nycomed Deutschland GmbH, Sprockhövel
  - Nycomed Deutschland GmbH, Stadthagen
  - Nycomed Deutschland GmbH, Starnberg
  - Nycomed Deutschland GmbH, Staudernheim
  - Nycomed Deutschland GmbH, Stavenhagen
  - Nycomed Deutschland GmbH, Steigra
  - Nycomed Deutschland GmbH, Steinen-Höllstein
  - Nycomed Deutschland GmbH, Steinfeld
  - Nycomed Deutschland GmbH, Steinwiesen
  - Nycomed Deutschland GmbH, Stendal
  - Nycomed Deutschland GmbH, Sternberg
  - Nycomed Deutschland GmbH, Stiege
  - Nycomed Deutschland GmbH, Stockelsdorf
  - Nycomed Deutschland GmbH, Stollberg
  - Nycomed Deutschland GmbH, Stolpen
  - Nycomed Deutschland GmbH, Straubing
  - Nycomed Deutschland GmbH, Strausberg
  - Nycomed Deutschland GmbH, Stuhr
  - Nycomed Deutschland GmbH, Stuttgart
  - Nycomed Deutschland GmbH, Stützengrün
  - Nycomed Deutschland GmbH, Suhl
  - Nycomed Deutschland GmbH, Sulingen
  - Nycomed Deutschland GmbH, Sulz-Glatt
  - Nycomed Deutschland GmbH, Sulzbach
  - Nycomed Deutschland GmbH, Sulzbach-Rosenberg
  - Nycomed Deutschland GmbH, Sulzfeld
  - Nycomed Deutschland GmbH, Sünna
  - Nycomed Deutschland GmbH, Tangerhütte
  - Nycomed Deutschland GmbH, Tangermünde
  - Nycomed Deutschland GmbH, Tarp
  - Nycomed Deutschland GmbH, Taucha
  - Nycomed Deutschland GmbH, Taunusstein
  - Nycomed Deutschland GmbH, Teltow
  - Nycomed Deutschland GmbH, Tessin
  - Nycomed Deutschland GmbH, Thum-Jahnsbach
  - Nycomed Deutschland GmbH, Thurnau
  - Nycomed Deutschland GmbH, Titz-Rödingen
  - Nycomed Deutschland GmbH, Torgelow
  - Nycomed Deutschland GmbH, Tönisvorst
  - Nycomed Deutschland GmbH, Trappenkamp
  - Nycomed Deutschland GmbH, Treffurt
  - Nycomed Deutschland GmbH, Triebes
  - Nycomed Deutschland GmbH, Triptis
  - Nycomed Deutschland GmbH, Trossingen
  - Nycomed Deutschland GmbH, Tutow
  - Nycomed Deutschland GmbH, Uelzen
  - Nycomed Deutschland GmbH, Uhlstädt
  - Nycomed Deutschland GmbH, Ulm
  - Nycomed Deutschland GmbH, Umkirch
  - Nycomed Deutschland GmbH, Unterhaching
  - Nycomed Deutschland GmbH, Unterschneidheim
  - Nycomed Deutschland GmbH, Unterwellenborn OT Goßwitz
  - Nycomed Deutschland GmbH, Urbach
  - Nycomed Deutschland GmbH, Uslar/Volpriehausen
  - Nycomed Deutschland GmbH, Vaihingen
  - Nycomed Deutschland GmbH, Vallendar
  - Nycomed Deutschland GmbH, Veilsdorf
  - Nycomed Deutschland GmbH, Velbert
  - Nycomed Deutschland GmbH, Vellahn
  - Nycomed Deutschland GmbH, Veringenstadt
  - Nycomed Deutschland GmbH, Vierkirchen
  - Nycomed Deutschland GmbH, Viersen
  - Nycomed Deutschland GmbH, Vilshofen
  - Nycomed Deutschland GmbH, Visselhövede
  - Nycomed Deutschland GmbH, Vitzenburg
  - Nycomed Deutschland GmbH, Voerde
  - Nycomed Deutschland GmbH, Völklingen
  - Nycomed Deutschland GmbH, VS-Schwenningen
  - Nycomed Deutschland GmbH, Wachau
  - Nycomed Deutschland GmbH, Wadern
  - Nycomed Deutschland GmbH, Wadgassen
  - Nycomed Deutschland GmbH, Waidhaus
  - Nycomed Deutschland GmbH, Waldbröl
  - Nycomed Deutschland GmbH, Waldbrunn-Strümpfelbrunn
  - Nycomed Deutschland GmbH, Wallwitz
  - Nycomed Deutschland GmbH, Walsleben
  - Nycomed Deutschland GmbH, Wandersleben
  - Nycomed Deutschland GmbH, Wanzleben
  - Nycomed Deutschland GmbH, Warin
  - Nycomed Deutschland GmbH, Warstein
  - Nycomed Deutschland GmbH, Wattenheim
  - Nycomed Deutschland GmbH, Wedel
  - Nycomed Deutschland GmbH, Wegberg
  - Nycomed Deutschland GmbH, Wegeleben
  - Nycomed Deutschland GmbH, Wehrsdorf
  - Nycomed Deutschland GmbH, Weibern
  - Nycomed Deutschland GmbH, Weida
  - Nycomed Deutschland GmbH, Weiden I.d. Oberpfalz
  - Nycomed Deutschland GmbH, Weiden i.d.Oberpfalz
  - Nycomed Deutschland GmbH, Weimar
  - Nycomed Deutschland GmbH, Weinböhla
  - Nycomed Deutschland GmbH, Weinheim-Oberflockenbach
  - Nycomed Deutschland GmbH, Weinsberg
  - Nycomed Deutschland GmbH, Weisenheim am Sand
  - Nycomed Deutschland GmbH, Weissensee
  - Nycomed Deutschland GmbH, Weißenburg
  - Nycomed Deutschland GmbH, Weißenfels
  - Nycomed Deutschland GmbH, Weißwasser
  - Nycomed Deutschland GmbH, Welden
  - Nycomed Deutschland GmbH, Welver
  - Nycomed Deutschland GmbH, Wennigsen
  - Nycomed Deutschland GmbH, Wernigerode
  - Nycomed Deutschland GmbH, Wesel
  - Nycomed Deutschland GmbH, Wesselburen
  - Nycomed Deutschland GmbH, Westerkappeln
  - Nycomed Deutschland GmbH, Westerrönfeld
  - Nycomed Deutschland GmbH, Westhausen
  - Nycomed Deutschland GmbH, Wettringen
  - Nycomed Deutschland GmbH, Wetzlar
  - Nycomed Deutschland GmbH, Wickede
  - Nycomed Deutschland GmbH, Wiehl
  - Nycomed Deutschland GmbH, Wiesbaden
  - Nycomed Deutschland GmbH, Wiesloch
  - Nycomed Deutschland GmbH, Wilburgstetten
  - Nycomed Deutschland GmbH, Wildeshausen
  - Nycomed Deutschland GmbH, Wilhelmsfeld
  - Nycomed Deutschland GmbH, Wilhelmshaven
  - Nycomed Deutschland GmbH, Willebadessen
  - Nycomed Deutschland GmbH, Willich
  - Nycomed Deutschland GmbH, Wilster
  - Nycomed Deutschland GmbH, Winkelhaid
  - Nycomed Deutschland GmbH, Winsen
  - Nycomed Deutschland GmbH, Wismar
  - Nycomed Deutschland GmbH, Witten
  - Nycomed Deutschland GmbH, Wittenberg
  - Nycomed Deutschland GmbH, Witzenhausen
  - Nycomed Deutschland GmbH, Wolfen
  - Nycomed Deutschland GmbH, Worbis
  - Nycomed Deutschland GmbH, Wörnitz
  - Nycomed Deutschland GmbH, Wörrstadt
  - Nycomed Deutschland GmbH, Wörth
  - Nycomed Deutschland GmbH, Wriedel
  - Nycomed Deutschland GmbH, Wulfen
  - Nycomed Deutschland GmbH, Wuppertal
  - Nycomed Deutschland GmbH, Wurzen
  - Nycomed Deutschland GmbH, Wustrau
  - Nycomed Deutschland GmbH, Wümbach
  - Nycomed Deutschland GmbH, Würzburg
  - Nycomed Deutschland GmbH, Zerbst
  - Nycomed Deutschland GmbH, Zittau
  - Nycomed Deutschland GmbH, Zittau-Wittgendorf
  - Nycomed Deutschland GmbH, Zorge
  - Nycomed Deutschland GmbH, Zossen
  - Nycomed Deutschland GmbH, Zschopau
  - Nycomed Deutschland GmbH, Zschorlau
  - Nycomed Deutschland GmbH, Zweibrücken
  - Nycomed Deutschland GmbH, Zwickau
  - Nycomed Deutschland GmbH, Zwönitz

RESULTS

PARTICIPANT FLOW:
Groups:
- Matrifen®: All patients enrolled
Period: Overall Study
Arm/Group | Matrifen®
Started | 5308
Completed | 5080
Not Completed | 228
Not completed — Combination of multiple reasons | 176
Not completed — Missing data | 52

BASELINE CHARACTERISTICS:
Arm/Group | Matrifen®
Number analyzed (Participants) | 5308
Age Continuous [Mean (Standard Deviation); unit: years] — The reported values are related to the number of 5174 subjects. This number differs from the overall number of baseline participants due to missing data for 134 subjects.
  years | 70.3 (13.2)
Gender [Number; unit: participants] — The reported values are related to the number of 5305 subjects. This number differs from the overall number of baseline participants due to missing data for 3 subjects.
  participants
    Female | 3334
    Male | 1971
Type of pain [Number; unit: participants] — Multiple types of pain possible. One participant can have more than one type of pain.
  participants
    Severe pain when moving | 3751
    Pain caused by a tumor | 1359
    Other type of pain | 877
    Missing data | 7
Underlying disease [Number; unit: Participants] — Multiple diseases possible. One participant can have more than one underlying disease.
  Participants
    Musculoskeletal disorders | 3396
    Tumor | 1416
    Neurological disorders | 514
    Dermatological disorders | 51
    Underlying disease NOS | 210
    Missing data | 371

OUTCOME MEASURES:

1. Primary Outcome: Patient's Assessment of Pain Severity Score
Description: Assessment on a Visual Analogue Scale from 0=No pain to 10=Most severe pain
Time Frame: Before and after therapy with Matrifen® (4 weeks)
Population: Patients included and treated with valid data at first and last visit (without imputation of missing values), intention to treat
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- Matrifen®: All patients with valid values at first and last visit
Arm/Group | Matrifen®
Number analyzed (Participants) | 5226
Units on a scale
  Start of therapy | 7.12 (1.52)
  End of study | 3.32 (1.66)

2. Primary Outcome: Physician's Final Assessment of the Efficacy of Therapy With Matrifen®
Description: Assessment on a scale: Excellent, good, satisfactory, dissatisfactory
Time Frame: After 4 week therapy with Matrifen®
Population: All patients included and treated, intention to treat, missing values not imputed
Measure: Number; unit: Participants
Groups:
- Matrifen®: All patients with valid values ('as observed')
Arm/Group | Matrifen®
Number analyzed (Participants) | 5308
Participants
  Excellent | 2530
  Good | 2273
  Satisfactory | 365
  Dissatisfactory | 73
  Missing data | 67

3. Primary Outcome: EQ-5D (Optional): Domain Mobility
Description: This outcome measure to assess patients quality of life is based on an optional standardised patient questionnaire (EQ-5D).
  Questions on a scale from 1-3 at initial and final visit:
  1. I have no problems in walking around
  2. I have some problems in walking around
  3. I am confined to bed
Time Frame: Before and after therapy with Matrifen® (4 weeks)
Population: as for outcome 1
Measure: Number; unit: Participants
Groups:
- Matrifen® / Initial Visit; Matrifen® / Final Visit: All patients with valid values at first and last visit
Arm/Group | Matrifen® / Initial Visit | Matrifen® / Final Visit
Number analyzed (Participants) | 3435 | 3435
Participants
  I have no problems in walking around | 284 | 1294
  I have some problems in walking around | 2779 | 1923
  I am confined to bed | 372 | 218

4. Primary Outcome: EQ-5D (Optional): Domain Mobility
Description: as for outcome 3
Time Frame: Before and after therapy with Matrifen® (4 weeks)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Matrifen® / Initial Visit | Matrifen® / Final Visit
Number analyzed (Participants) | 3435 | 3435
Units on a scale | 2.03 (0.44) | 1.69 (0.58)

5. Primary Outcome: EQ-5D (Optional): Domain Self Care
Description: This outcome measure to assess patients quality of life is based on an optional standardised patient questionnaire (EQ-5D).
  Questions on a scale from 1-3 at initial and final visit:
  1. I have no problems with self-care
  2. I have some problems washing or dressing myself
  3. I am unable to wash or dress myself
Time Frame: Before and after therapy with Matrifen® (4 weeks)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Matrifen® / Initial Visit | Matrifen® / Final Visit
Number analyzed (Participants) | 3435 | 3435
Participants
  I have no problems with self-care | 682 | 1709
  I have some problems washing or dressing myself | 2152 | 1461
  I am unable to wash or dress myself | 601 | 265

6. Primary Outcome: EQ-5D (Optional): Domain Self Care
Description: as for outcome 5
Time Frame: Before and after therapy with Matrifen® (4 weeks)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Matrifen® / Initial Visit | Matrifen® / Final Visit
Number analyzed (Participants) | 3435 | 3435
Units on a scale | 1.98 (0.61) | 1.58 (0.63)

7. Primary Outcome: EQ-5D (Optional): Domain Usual Activities
Description: This outcome measure to assess patients quality of life is based on an optional standardised patient questionnaire (EQ-5D).
  Questions on a scale from 1-3 at initial and final visit:
  1. I have no problems with performing my usual activities
  2. I have some problems with performing my usual activities
  3. I am unable to perform my usual activities
Time Frame: Before and after therapy with Matrifen® (4 weeks)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Matrifen® / Initial Visit | Matrifen® / Final Visit
Number analyzed (Participants) | 3435 | 3435
Participants
  I have no problems with performing my usual activi | 142 | 1070
  I have some problems with performing my usual acti | 2227 | 1973
  I am unable to perform my usual activities | 1066 | 392

8. Primary Outcome: EQ-5D (Optional): Domain Usual Activities
Description: as for outcome 7
Time Frame: Before and after therapy with Matrifen® (4 weeks)
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Matrifen® / Initial Visit | Matrifen® / Final Visit
Number analyzed (Participants) | 3435 | 3435
Units on a scale | 2.27 (0.53) | 1.80 (0.62)

9. Primary Outcome: EQ-5D (Optional): Pain / Discomfort
Description: This outcome measure to assess patients quality of life is based on an optional standardised patient questionnaire (EQ-5D).
  Questions on a scale from 1-3 at initial and final visit:
  1. I have no pain or discomfort
  2. I have moderate pain or discomfort
  3. I have extreme pain or discomfort
Time Frame: Before and after therapy with Matrifen® (4 weeks)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Matrifen® / Initial Visit | Matrifen® / Final Visit
Number analyzed (Participants) | 3435 | 3435
Participants
  I have no pain or discomfort | 18 | 749
  I have moderate pain or discomfort | 1104 | 2503
  I have extreme pain or discomfort | 2313 | 183

10. Primary Outcome: EQ-5D (Optional): Pain / Discomfort
Description: as for outcome 9
Time Frame: Before and after therapy with Matrifen® (4 weeks)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Matrifen® / Initial Visit | Matrifen® / Final Visit
Number analyzed (Participants) | 3435 | 3435
Units on a scale | 2.67 (0.48) | 1.84 (0.49)

11. Secondary Outcome: Physician's Assessment of the Skin Tolerability of the Fentanyl-patches
Description: Assessment on a scale: Excellent, good, satisfactory, dissatisfactory
Time Frame: After 4 week therapy with Matrifen®
Population: All patients included and treated, intention to treat, missing values not imputed
Measure: Number; unit: Participants
Arm/Group | Matrifen®
Number analyzed (Participants) | 5308
Participants
  Excellent | 3403
  Good | 1716
  Satisfactory | 82
  Dissatisfactory | 18
  Missing data | 89

12. Secondary Outcome: Patient's Assessment of the Acceptance of the Fentanyl-patches
Description: Assessment on a scale: Excellent, good, satisfactory, dissatisfactory
Time Frame: After 4 week therapy with Matrifen®
Population: All patients included and treated, intention to treat, missing values not imputed
Measure: Number; unit: Participants
Arm/Group | Matrifen®
Number analyzed (Participants) | 5308
Participants
  Excellent | 3210
  Good | 1725
  Satisfactory | 168
  Dissatisfactory | 101
  Missing data | 104

13. Primary Outcome: EQ-5D (Optional): Domain Anxiety / Depression
Description: This outcome measure to assess patients quality of life is based on an optional standardised patient questionnaire (EQ-5D).
  Questions on a scale from 1-3 at initial and final visit:
  1. I am not anxious or depressed
  2. I am moderately anxious or depressed
  3. I am extremely anxious or depressed
Time Frame: Before and after therapy with Matrifen® (4 weeks)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Matrifen® / Initial Visit | Matrifen® / Final Visit
Number analyzed (Participants) | 3435 | 3435
Participants
  I am not anxious or depressed | 688 | 1920
  I am moderately anxious or depressed | 1949 | 1409
  I am extremely anxious or depressed | 798 | 106

14. Primary Outcome: EQ-5D (Optional): Domain Anxiety / Depression
Description: as for outcome 13
Time Frame: Before and after therapy with Matrifen® (4 weeks)
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Matrifen® / Initial Visit | Matrifen® / Final Visit
Number analyzed (Participants) | 3435 | 3435
Units on a scale | 2.03 (0.66) | 1.47 (0.56)

15. Primary Outcome: EQ-5D (Optional): European Index Score
Description: Index derived from the five EQ-5D-items (= mobility, self care, usual activities, pain/discomfort, anxiety/depression) resulting in a value from -1= very ill to 1=full health
Time Frame: Before and after therapy with Matrifen® (4 weeks)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Matrifen®
Number analyzed (Participants) | 3435
Units on a scale
  Initial visit | 0.078 (0.35)
  Final visit | 0.584 (0.31)

16. Primary Outcome: EQ-5D (Optional): Visual Analogue Scale
Description: Visual Analogue Scale (VAS) from 0 =worst imaginable health status, 100 =best imaginable health status
Time Frame: Before and after therapy with Matrifen® (4 weeks)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Matrifen®
Number analyzed (Participants) | 3435
Units on a scale
  Initial visit | 40.1 (22.0)
  Final visit | 58.8 (20.4)

17. Secondary Outcome: Physician's Assessment of the Adhesion Properties of the Fentanyl-patches
Description: Assessment on a scale: Excellent, good, satisfactory, dissatisfactory
Time Frame: After 4 week therapy with Matrifen®
Population: All patients included and treated, intention to treat, missing values not imputed
Measure: Number; unit: Participants
Arm/Group | Matrifen®
Number analyzed (Participants) | 5308
Participants
  Excellent | 3274
  Good | 1777
  Satisfactory | 162
  Dissatisfactory | 35
  Missing data | 60

18. Secondary Outcome: Physician's Final Assessment of the Tolerability of Matrifen®
Description: Assessment on a scale: Excellent, good, satisfactory, dissatisfactory
Time Frame: After 4 week therapy with Matrifen®
Population: All patients included and treated, intention to treat, missing values not imputed
Measure: Number; unit: Participants
Arm/Group | Matrifen®
Number analyzed (Participants) | 5308
Participants
  Excellent | 2866
  Good | 2058
  Satisfactory | 161
  Dissatisfactory | 75
  Missing data | 148

ADVERSE EVENTS:
Time Frame: First until last visit (planned: 4 weeks)
Groups:
- Matrifen®: Patients included and treated with at least one application of Matrifen®
Arm/Group | Matrifen®
Serious Adverse Events (participants affected / at risk) | 80/5308
Other Adverse Events (participants affected / at risk) | 0/5308
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Matrifen® (N=5308)
Cardiac failure (Cardiac disorders) | 1 (1)
Cardiovascular disorder (Cardiac disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 1 (1)
Death (General disorders) | 49 (49)
General physical health deterioration (General disorders) | 1 (1)
Metastases to liver (Hepatobiliary disorders) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Pelvic fracture (Injury, poisoning and procedural complications) | 1 (1)
Metastases to bone (Musculoskeletal and connective tissue disorders) | 1 (1)
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Dementia Alzheimer's type (Psychiatric disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1)
Hospitalisation (Surgical and medical procedures) | 14 (14)
Surgery (Surgical and medical procedures) | 6 (6)
Amputation (Surgical and medical procedures) | 1 (1)
Prosthesis implantation (Surgical and medical procedures) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No